CLINICAL TRIAL: NCT06092996
Title: Sling vs No Sling After Reverse Total Shoulder Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00113901
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Disease; Rotator Cuff Tear Arthropathy; Shoulder Osteoarthritis
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling (No Intervention): Participants in the sling group will wear a sling according to current standard of care: 3 weeks postoperatively (2 weeks all the time, 3rd week at night and while in the community)
- No Sling (Experimental): Participants in the no sling group will only wear a sling for three days postoperatively
  Interventions: Other: Time of Sling Use

INTERVENTIONS:
Other: Time of Sling Use — Standard sling worn for only three days post operatively
  Arms: No Sling

SUMMARY:
This study involves patients who will be undergoing a reverse total shoulder replacement at Duke University. 100 eligible will be randomly assigned into one of two groups, a sling or no sling group. Patients in the sling group will wear a sling for three weeks after their surgery while the no sling group will only wear a sling three days after their surgery. Patients will follow their doctors normal follow up visit schedule after surgery, with visits at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether or not a sling is necessary after the nerve block has worn off postoperatively for patients undergoing reverse total shoulder arthroplasty. Patients who are scheduled for a reverse total shoulder with the participating investigators will be approached for potential participation in the study.

Before the surgery, subjects will be randomly assigned to either the Sling (control) group or the No-Sling (investigational) group. The Sling, or control, group will wear a sling through 3 weeks postoperatively. The No Sling (investigational) group, will wear a sling either through 3 days postoperatively.

Following surgery, patients will be followed at their standard of care visits at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after their surgical date. The investigators will collect data from these standard of care visits including PROs (including but not limited to ASES and SANE), Adverse events data, and physical exam data including range of motion. Patients will be followed through their two-year visit and then taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo a primary reverse shoulder arthroplasty procedure
* Patient voluntarily consents to participate in the study and has the mental and physical ability to participate in the study, fill out subjective questionnaires, return for follow-up visits, and comply with prescribed post-operative physical therapy
* Patient meets indications for primary reverse shoulder arthroplasty for the following diagnosis
* Rotator cuff arthropathy
* Glenohumeral arthritis
* Patient is between 18-100 years old
* Patient is English speaking

Exclusion Criteria:

* A history of ipsilateral shoulder arthroplasty
* A history of shoulder septic arthritis
* A history of a proximal humeral fracture
* Chronic locked dislocation
* Rheumatoid arthritis
* Tumors
* Axillary nerve damage
* Non-functioning deltoid muscle
* Glenoid vault deficiency precluding baseplate fixation
* Infection and neuropathic joints
* Known or suspected non-compliance, drug or alcohol abuse
* Patients incapable of judgement or under tutelage
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, contraindication for imaging etc.
* The subject is related to investigator as family members, employees, or other dependent persons

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop any kind of postoperative complication | 6 months primary, Up to the first 2 years following surgery
  Incidence of postoperative complications

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) score | 6 months primary, Up to the first 2 years following surgery
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. Total score ranges from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Single Assessment Numeric Evaluation (SANE) score | 6 months primary, Up to the first 2 years following surgery
  The SANE is a single-question outcome measure that asks patients to rate their function (as it pertains to the area being treated) on a scale of 0 to 100, where a higher score indicates greater function.

CONTACTS AND LOCATIONS:
Overall Officials: Oke A Anakwenze, MD, MBA, Principal Investigator — Duke University; Christopher Klifto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No